CLINICAL TRIAL: NCT01755013
Title: Open-label Observational Study of Plastic Cylindrical Fiber Optic Diffuser (Pioneer Optics) in Photodynamic Therapy for the Management of Cholangiocarcinoma.
Brief Title: Photodynamic Therapy (PDT) for Palliation of Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief of Advanced Endoscopy, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1110011999
Record Dates: First submitted 2012-03-01; First posted 2012-12-21 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Cholangiocarcinoma; Biliary Stricture; Biliary Obstruction; Bile Duct Cancer
Keywords: Cholangiocarcinoma; Biliary Stricture; Biliary obstruction; Bile Duct Cancer; PDT; Photodynamic Therapy; Plastic optic Diffuser; Laser
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDT Group (Experimental): Subjects who receive Photodynamic therapy with plastic optic diffuser.
  Interventions: Procedure: Photodynamic Therapy

INTERVENTIONS:
Procedure: Photodynamic Therapy — Photofrin and Photodynamic therapy using the plastic optic diffuser, conducted during Standard of care Endoscopic retrograde cholangiopancreatography (ERCP)
  Other Names: PDT; Laser

SUMMARY:
Successful palliation of biliary obstruction is the main goal for reducing morbidity and mortality in patients with biliary disease and biliary obstruction related to cholangiocarcinoma. Surgical intervention for the sale is unfortunately complicated by a 30-day postoperative mortality rate of between 7 and 24%. Moreover, because of recovery time the quality of life following surgery is only improved in a minority. At present endoscopic insertion of a plastic or metal stent is the method of choice to relieve obstructive jaundice without the high morbidity and mortality associated with surgery. But this relief is unfortunately temporary since stents tend to become obstructed and the fact that effective biliary drainage in the proximal lesion is challenging.

Photodynamic Therapy (PDT) is a new therapeutic approach that specifically targets neoplastic cells. This therapy involves the intravenous administration of a photosensitizing agent followed by activation of the agent by illumination with non-thermal light of a specific wavelength, resulting in cell death from direct cytotoxicity and ischemic necrosis. A randomized controlled trial study by Ortner et all confirmed the significant advantage of PDT with regard to relief of jaundice, quality of life, and survival.

In photodynamic therapy (PDT) the uniform distribution of externally applied light is desirable but often difficult to achieve. An optical fiber tip producing cylindrical or lateral light emission can facilitate the application of laser energy by direct implantation of the tip into solid tumors. However, currently used FDA approved glass diffusers used in standard of care PDT might break in the bile ducts causing injury since they are not meant to be used within bile ducts through an endoscope or choledochoscope. Hence, there is a need to evaluate and introduce more efficient and safe non-glass cylindrical optic fiber diffuser for photo dynamic therapy in the bile ducts. Recent studies have shown that the Pioneer plastic optic diffuser is safe and effective in photodynamic therapy, it can be also used via a choledochoscope. We aim to add to the clinical evidence by conducting an open label observational study trial using this fiber optic diffuser during photo dynamic therapy in the bile ducts.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is the second most common malignancy arising within the liver, and the association of this malignant condition with high morbidity and mortality is well recognized. It originates from the epithelium of bile ducts or ductules. Two types have been described: the peripheral type occurring in the parenchyma of the liver and the central type occurring within or related to the major bile ducts. Surgery can offer a curative chance, but only a minority of patients are candidates for this therapy at initial presentation since most patients are found with an unresectable tumor.

In unresectable cases, the median survival is 6 months. Since morbidity and mortality from CCA occurs because of biliary obstruction, successful palliation of that complication is the main goal in these patients. Surgical biliary bypass can be offered in order to prolong life and relieve symptoms. This intervention is unfortunately complicated by 30-day postoperative mortality rate between 7 and 24%. Moreover, the quality of life following surgery is only improved in a minority because of the time needed to recover from surgery.

Endoscopic biliary stenting during endoscopic retrograde cholangiopancreatography (ERCP) offers relief from obstructive jaundice without the high morbidity and mortality associated with surgery. In addition, a study by Luman et al even showed significant improvement in emotional, cognitive and global health scores following stenting. But this relief is unfortunately temporary since stents tend to become obstructed.

Local therapies including iridium brachytherapy and photodynamic therapy (PDT) may prevent or postpone these problems.

For more information about PDT, please see the 'Citations' section.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cholangiocarcinoma
* Patient is age 18 years or older
* Patient is receiving Photodynamic therapy with stent(s) placement as part of their original treatment plan
* Patients must have adequate coagulation as defined below:

Patient's INR ≤ 2 within 30 days of treatment Patient's platelets > 50,000/cmm within 30 days of treatment

Exclusion Criteria:

* Subject has acute porphyria. Subjects exhibiting neurologic or cutaneous symptoms will undergo urinary delta-aminolevulinic acid and porphobilinogen dosage tests to determine severity.
* Subject is pregnant.
* Subject is allergic to Photofrin.
* Subject has uncorrected coagulopathy
* Subject is unstable for ERCP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-01-22 (Estimated); Study Completion 2018-03-22 (Estimated)

PRIMARY OUTCOMES:
Efficacy Profile | 2 months
  To assess the efficacy of a plastic cylindrical fiber optic diffuser (Pioneer Optics) in photodynamic therapy for the management of Cholangiocarcinoma by visualization of visible necrosis of target tissue in bile ducts after the application of the device.

SECONDARY OUTCOMES:
Safety Profile | 2 months
  To assess the the number and intensity of adverse events occurring due to the application of the research device.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD

REFERENCES:
- [Background] Talreja JP, DeGaetani M, Sauer BG, Kahaleh M. Photodynamic therapy for unresectable cholangiocarcinoma: contribution of single operator cholangioscopy for targeted treatment. Photochem Photobiol Sci. 2011 Jul;10(7):1233-8. doi: 10.1039/c0pp00259c. Epub 2011 Apr 21. PMID 21512706
- [Background] Richter JA, Kahaleh M. Photodynamic therapy: Palliation and endoscopic technique in cholangiocarcinoma. World J Gastrointest Endosc. 2010 Nov 16;2(11):357-61. doi: 10.4253/wjge.v2.i11.357. PMID 21173912
- [Background] Talreja JP, Kahaleh M. Photodynamic therapy for cholangiocarcinoma. Gut Liver. 2010 Sep;4 Suppl 1(Suppl 1):S62-6. doi: 10.5009/gnl.2010.4.S1.S62. Epub 2010 Sep 10. PMID 21103297
- See also: Photodynamic therapy for unresectable cholangiocarcinoma: contribution of single operator cholangioscopy for targeted treatment. Talreja JP, DeGaetani M, Sauer BG, Kahaleh M. — http://www.ncbi.nlm.nih.gov/pubmed/21512706
- See also: Photodynamic therapy: Palliation and endoscopic technique in cholangiocarcinoma. Richter JA, Kahaleh M. — http://www.ncbi.nlm.nih.gov/pubmed/21173912
- See also: Photodynamic therapy for cholangiocarcinoma. Talreja JP, Kahaleh M. — http://www.ncbi.nlm.nih.gov/pubmed/21103297